CLINICAL TRIAL: NCT05475158
Title: Comparison of Optical Coherence Tomography Angiographic Factors of Macula and Optic Disc in Patients With or Without Amyloid Pathology: A Prospective Study
Brief Title: Comparison of OCTA Factors in Patients With or Without Amyloid Pathology: A Prospective Study
Status: Completed | Type: Observational
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1908-004-081
Record Dates: First submitted 2022-06-23; First posted 2022-07-26 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Alzheimer Disease; Amyloid Angiopathy; Macular Ischemia; Dementia; Mild Cognitive Impairment
Keywords: Alzheimer disease dementia; Mild cognitive impairment; Amyloid pathology; Optical coherence tomographic angiography
MeSH Terms: conditions — Alzheimer Disease; Amyloid angiopathy; Dementia; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Dementia: Patients with Alzheimer disease dementia (ADD) fulfilled the NIA-AA core clinical criteria for probable ADD and Aβ positive according to ATN classification scheme.
  Aβ positive refers to Aβ pathology (CSF Aβ1-42 < 631.8 pg/ml or positive amyloid deposits on 18F-flutemetamol PET by visual inspection).
- MCI (Mild cognitive impairment): Patients with mild cognitive impairment (MCI) met the Petersen's criteria.
- CU (Cognitively unimpaired control): CU consisted of cognitively unimpaired subjects whose cognition (as defined by the Seoul Neuropsychological Screening Battery (SNSB)) was within normal limits.
- Aβ positive: Aβ positive refers to Aβ pathology (CSF Aβ1-42 < 631.8 pg/ml or positive amyloid deposits on 18F-flutemetamol PET by visual inspection).
- Aβ negative: Aβ negative was within normal limits.

SUMMARY:
To compare alternation of retinal microcirculation within the macula and optic disc in patients with dementia, mild cognitive impairment (MCI), and cognitively healthy subjects who had positive amyloid biomarkers (Aβ +) or not, using optical coherence tomography angiography (OCTA).

DETAILED DESCRIPTION:
Alzheimer disease dementia (ADD) is the most common neurodegenerative disease dementia in elderly population associated with the accumulation of beta-amyloid (Aβ) plaques and tau neurofibrillary tangles (NFTs). Diagnostic biomarkers reflecting underlying amyloid or tau pathology of ADD have actively been developed. Of these, amyloid or tau positron emission tomography (PET) imaging and cerebrospinal fluid (CSF) Aβ1-42 or phosphorylated tau are representative biomarkers for ADD. However, these tend to be expensive, invasive, or available only in a tertiary hospital or a specialized laboratory. Alternative biomarkers which are inexpensive, less invasive, and highly available could be needed.

Patients with ADD commonly show visuospatial dysfunction which is mainly attributed to damage of parieto-occipital or temporo-occipital visual pathway. In addition, previous studies using optical coherence tomography (OCT) which is a useful tool measuring retinal nerve fiber layer thickness (RNFLT), macula ganglion cell/inner plexiform layer thickness (GC/IPLT) reported impaired pregeniculate afferent visual pathway, for example, reduction of RNFLT and loss of retinal ganglionic cells (RGCs) in patients with ADD.

The retina and brain have the same embryological origin. These were branched off from the forebrain, so the brain and retina have similar anatomic and physiologic traits of the vasculature. In line with this, several studies using laser doppler ultrasonography, or retinal function imager (RFI) revealed narrowed central retinal vein and decreased its blood velocity, or low blood flow rate of retinal arterioles and venules in patients with mild cognitive impairment (MCI) and ADD. The authors suggested that in patients with ADD, accumulation of Aβ in the vessel walls could cause disruption of basement membrane and endothelium, leading to the decreased vascular lumen and density of retinal vessel. Indeed, postmortem study revealed accumulated Aβ inside or around RGCs in AD.

OCTA can clearly visualize not only the specific layers of retinal vasculatures, including superficial, middle, and deep capillary plexuses, but also choroidal vessels with a high resolution and in a reproducible manner, without contrast agent. A few prior studies using OCTA reported enlarged foveal avascular zone (FAZ) and decrease of retinal vascular density and choroidal thickness in ADD or MCI compared to controls. On the other hand, the others showed no differences in FAZ area and vessel density between them.

In this study, the investigators first evaluated structural and microvascular changes of retina and the microvascular change of macula and optic disc in patients with clinically diagnosed ADD, MCI and cognitively normal controls using OCT and OCTA. Then, to investigate whether impaired pregeniculate visual pathway is truly associated with underlying amyloid pathology, the investigators further investigated those OCT and OCTA parameters in each subgroup with positive or negative amyloid biomarker.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and pathologic diagnosis of ADD or MCI as well as cognitively unimpaired control (CU) from the Neurologic Clinic of Pusan National University Hospital

Exclusion Criteria:

* Patient not within the ages of 50-90 years old
* Patient with glaucoma, macular degeneration, retinal vascular disease including diabetic retinopathy, retinal vein occlusion
* Intraocular pressure (IOP) ≥ 21 mmHg
* Dense corneal or ocular media opacity
* History of ocular trauma or associated ocular disease
* Astigmatism ≥ 3.0 diopter or spherical equivalent ≥ 6.0 diopter
* Best corrected visual acuity (BCVA) < 20/40
* Any ocular surgery except uncomplicated cataract extraction
* Uncontrolled hypertension and diabetes

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neurologic Clinic of Pusan National University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
SD-OCT imaging | Through study completion, measured at enrollment and analyzed from September 2019 to July 2021
  Measuring macular GC/IPLT (μm) and cimcumpapillary RNFLT (μm).
  The average, minimum, and 6 sectoral (superotemporal, superior, superonasal, inferonasal, inferior, and inferotemporal) GC/IPLT (μm) values are obtained.
  The average, 4 sectoral (temporal, superior, nasal, and inferior), and 12 clock-hour circumpapillary RNFLT (μm) are obtained.
  Multiple measurements will not be aggregated, but analyzed respectively.
SD-OCTA imaging | Through study completion, measured at enrollment and analyzed from September 2019 to July 2021
  Acquiring microvasculature images of macular (6 × 6 mm^2 scan) and optic disc areas (4.5 × 4.5 mm^2 scan).
  The average vessel density (VD, mm/mm^2) and perfusion density (PD, %) were automatically measured in the Early Treatment of Diabetic Retinopathy Study (ETDRS) grid with values shown in the nine subfields, central, inner, outer and full region.
  The software calculated the area (mm^2), perimeter (mm), and circularity (defined as 4πA/P^2, where A was the area and P was the perimeter) of foveal avascular zone (FAZ). A circularity closer to 0 means an irregular shape, and closure to 1 indicates a circular shape.
  Multiple measurements will not be aggregated, but analyzed respectively.

SECONDARY OUTCOMES:
Diagnostic performance | Through study completion, analyzed from July 2021 to July 2022
  Diagnostic performance of OCT and OCTA parameters according to underlying Aβpathology.
  Receiver operating characteristic (ROC) curves were drawn by plotting sensitivity against 1-specificity, and areas under ROC curves (AUCs) were used to evaluate the diagnostic performance of continuous OCT/OCTA variables. Ideal cut-off points were derived using the Youden index
Correlations | Through study completion, analyzed from July 2021 to July 2022
  Correlations between MMSE score and all of OCT/OCTA parameters were expressed as Pearson's or Spearman's rank correlation coefficients to account for the normal or non-normal distribution of the parameters, respectively.
  OCT/OCTA parameters including as follows;
  1. macular GC/IPLT (μm): average, minimum, and 6 sectoral (superotemporal, superior, superonasal, inferonasal, inferior, and inferotemporal) GC/IPLT
  2. cimcumpapillary RNFLT (μm): verage, 4 sectoral (temporal, superior, nasal, and inferior), and 12 clock-hour circumpapillary RNFLT
  3. Macular vessel density (VD, mm/mm^2) & perfusion density (PD, %)
     : VDs and PDs of central, parafoveal (nasal, temporal, superior, inferior), perifoveal (nasal, temporal, superior, inferior), and total
  4. Optic disc perfusion density (%) and flux index (from 0 to 1) : nasal, temporal, superior, inferior

CONTACTS AND LOCATIONS:
Overall Officials: Eun-Joo Kim, MD, PhD, Principal Investigator — Department of Neurology, Pusan National University Hospital
Locations (1):
- Pusan National University Hospital, Busan, South Korea

REFERENCES:
- [Background] Arvanitakis Z, Shah RC, Bennett DA. Diagnosis and Management of Dementia: Review. JAMA. 2019 Oct 22;322(16):1589-1599. doi: 10.1001/jama.2019.4782. PMID 31638686
- [Background] Villemagne VL, Burnham S, Bourgeat P, Brown B, Ellis KA, Salvado O, Szoeke C, Macaulay SL, Martins R, Maruff P, Ames D, Rowe CC, Masters CL; Australian Imaging Biomarkers and Lifestyle (AIBL) Research Group. Amyloid beta deposition, neurodegeneration, and cognitive decline in sporadic Alzheimer's disease: a prospective cohort study. Lancet Neurol. 2013 Apr;12(4):357-67. doi: 10.1016/S1474-4422(13)70044-9. Epub 2013 Mar 8. PMID 23477989
- [Background] Clark CM, Pontecorvo MJ, Beach TG, Bedell BJ, Coleman RE, Doraiswamy PM, Fleisher AS, Reiman EM, Sabbagh MN, Sadowsky CH, Schneider JA, Arora A, Carpenter AP, Flitter ML, Joshi AD, Krautkramer MJ, Lu M, Mintun MA, Skovronsky DM; AV-45-A16 Study Group. Cerebral PET with florbetapir compared with neuropathology at autopsy for detection of neuritic amyloid-beta plaques: a prospective cohort study. Lancet Neurol. 2012 Aug;11(8):669-78. doi: 10.1016/S1474-4422(12)70142-4. Epub 2012 Jun 28. Erratum In: Lancet Neurol. 2012 Aug;11(8):658. PMID 22749065
- [Background] Albert MS, DeKosky ST, Dickson D, Dubois B, Feldman HH, Fox NC, Gamst A, Holtzman DM, Jagust WJ, Petersen RC, Snyder PJ, Carrillo MC, Thies B, Phelps CH. The diagnosis of mild cognitive impairment due to Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):270-9. doi: 10.1016/j.jalz.2011.03.008. Epub 2011 Apr 21. PMID 21514249
- [Background] Grossman I, Lutz MW, Crenshaw DG, Saunders AM, Burns DK, Roses AD. Alzheimer's disease: diagnostics, prognostics and the road to prevention. EPMA J. 2010 Jun;1(2):293-303. doi: 10.1007/s13167-010-0024-3. Epub 2010 Jun 29. PMID 21124753
- [Background] Kirby E, Bandelow S, Hogervorst E. Visual impairment in Alzheimer's disease: a critical review. J Alzheimers Dis. 2010;21(1):15-34. doi: 10.3233/JAD-2010-080785. PMID 20182034
- [Background] Hodges JR. Alzheimer's centennial legacy: origins, landmarks and the current status of knowledge concerning cognitive aspects. Brain. 2006 Nov;129(Pt 11):2811-22. doi: 10.1093/brain/awl275. PMID 17071920
- [Background] Cronin-Golomb A, Corkin S, Rizzo JF, Cohen J, Growdon JH, Banks KS. Visual dysfunction in Alzheimer's disease: relation to normal aging. Ann Neurol. 1991 Jan;29(1):41-52. doi: 10.1002/ana.410290110. PMID 1996878
- [Background] Blanks JC, Hinton DR, Sadun AA, Miller CA. Retinal ganglion cell degeneration in Alzheimer's disease. Brain Res. 1989 Nov 6;501(2):364-72. doi: 10.1016/0006-8993(89)90653-7. PMID 2819446
- [Background] Sadun AA, Bassi CJ. Optic nerve damage in Alzheimer's disease. Ophthalmology. 1990 Jan;97(1):9-17. doi: 10.1016/s0161-6420(90)32621-0. PMID 2314849
- [Background] Jiang H, Liu Y, Wei Y, Shi Y, Wright CB, Sun X, Rundek T, Baumel BS, Landman J, Wang J. Impaired retinal microcirculation in patients with Alzheimer's disease. PLoS One. 2018 Feb 2;13(2):e0192154. doi: 10.1371/journal.pone.0192154. eCollection 2018. PMID 29394263
- [Background] Brown WR, Thore CR. Review: cerebral microvascular pathology in ageing and neurodegeneration. Neuropathol Appl Neurobiol. 2011 Feb;37(1):56-74. doi: 10.1111/j.1365-2990.2010.01139.x. PMID 20946471
- [Background] Feke GT, Hyman BT, Stern RA, Pasquale LR. Retinal blood flow in mild cognitive impairment and Alzheimer's disease. Alzheimers Dement (Amst). 2015 Apr 23;1(2):144-51. doi: 10.1016/j.dadm.2015.01.004. eCollection 2015 Jun. PMID 27239502
- [Background] Berisha F, Feke GT, Trempe CL, McMeel JW, Schepens CL. Retinal abnormalities in early Alzheimer's disease. Invest Ophthalmol Vis Sci. 2007 May;48(5):2285-9. doi: 10.1167/iovs.06-1029. PMID 17460292
- [Background] Wu J, Zhang X, Azhati G, Li T, Xu G, Liu F. Retinal microvascular attenuation in mental cognitive impairment and Alzheimer's disease by optical coherence tomography angiography. Acta Ophthalmol. 2020 Sep;98(6):e781-e787. doi: 10.1111/aos.14381. Epub 2020 Mar 9. PMID 32153141
- [Background] Rosenfeld PJ, Durbin MK, Roisman L, Zheng F, Miller A, Robbins G, Schaal KB, Gregori G. ZEISS Angioplex Spectral Domain Optical Coherence Tomography Angiography: Technical Aspects. Dev Ophthalmol. 2016;56:18-29. doi: 10.1159/000442773. Epub 2016 Mar 15. PMID 27023249
- [Background] Nesper PL, Fawzi AA. Human Parafoveal Capillary Vascular Anatomy and Connectivity Revealed by Optical Coherence Tomography Angiography. Invest Ophthalmol Vis Sci. 2018 Aug 1;59(10):3858-3867. doi: 10.1167/iovs.18-24710. PMID 30073360
- [Background] de Carlo TE, Bonini Filho MA, Chin AT, Adhi M, Ferrara D, Baumal CR, Witkin AJ, Reichel E, Duker JS, Waheed NK. Spectral-domain optical coherence tomography angiography of choroidal neovascularization. Ophthalmology. 2015 Jun;122(6):1228-38. doi: 10.1016/j.ophtha.2015.01.029. Epub 2015 Mar 17. PMID 25795476
- [Background] Bulut M, Kurtulus F, Gozkaya O, Erol MK, Cengiz A, Akidan M, Yaman A. Evaluation of optical coherence tomography angiographic findings in Alzheimer's type dementia. Br J Ophthalmol. 2018 Feb;102(2):233-237. doi: 10.1136/bjophthalmol-2017-310476. Epub 2017 Jun 9. PMID 28600299
- [Background] Jiang H, Wei Y, Shi Y, Wright CB, Sun X, Gregori G, Zheng F, Vanner EA, Lam BL, Rundek T, Wang J. Altered Macular Microvasculature in Mild Cognitive Impairment and Alzheimer Disease. J Neuroophthalmol. 2018 Sep;38(3):292-298. doi: 10.1097/WNO.0000000000000580. PMID 29040211
- [Background] O'Bryhim BE, Apte RS, Kung N, Coble D, Van Stavern GP. Association of Preclinical Alzheimer Disease With Optical Coherence Tomographic Angiography Findings. JAMA Ophthalmol. 2018 Nov 1;136(11):1242-1248. doi: 10.1001/jamaophthalmol.2018.3556. PMID 30352114
- [Background] Zhang YS, Zhou N, Knoll BM, Samra S, Ward MR, Weintraub S, Fawzi AA. Parafoveal vessel loss and correlation between peripapillary vessel density and cognitive performance in amnestic mild cognitive impairment and early Alzheimer's Disease on optical coherence tomography angiography. PLoS One. 2019 Apr 2;14(4):e0214685. doi: 10.1371/journal.pone.0214685. eCollection 2019. PMID 30939178
- [Background] den Haan J, van de Kreeke JA, van Berckel BN, Barkhof F, Teunissen CE, Scheltens P, Verbraak FD, Bouwman FH. Is retinal vasculature a biomarker in amyloid proven Alzheimer's disease? Alzheimers Dement (Amst). 2019 May 10;11:383-391. doi: 10.1016/j.dadm.2019.03.006. eCollection 2019 Dec. PMID 31193094
- [Background] van de Kreeke JA, Nguyen HT, Konijnenberg E, Tomassen J, den Braber A, Ten Kate M, Yaqub M, van Berckel B, Lammertsma AA, Boomsma DI, Tan SH, Verbraak F, Visser PJ. Optical coherence tomography angiography in preclinical Alzheimer's disease. Br J Ophthalmol. 2020 Feb;104(2):157-161. doi: 10.1136/bjophthalmol-2019-314127. Epub 2019 May 22. PMID 31118186